CLINICAL TRIAL: NCT02187250
Title: Short-term Treatment With PDE-4 Inhibitor Roflumilast or GLP-1 Agonist Liraglutide or Metformin in Treatment Naive Obese Women With Polycystic Ovary Syndrome
Brief Title: PDE-4 Inhibitor Roflumilast and GLP-1 Agonist Liraglutide in Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, professor, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAXAS 2
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: PCOS; Obesity
Keywords: PCOS; PDE-4 inhibitor; roflumilast; liraglutide; metformin; obesity
MeSH Terms: conditions — Obesity | interventions — Metformin; Liraglutide; Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- metformin (Active Comparator): In the metformin group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 2x1000 mg BID per os.
  Interventions: Drug: metformin
- liraglutide (Active Comparator): In the liraglutide group liraglutide was initiated at a dose of 0,6mg sc once per day for one week and increased to 1,2mg sc one per day.
  Interventions: Drug: liraglutide
- roflumilast (Active Comparator): In the roflumilast group roflumilast was initiated at a dose of 500 mg BID per os.
  Interventions: Drug: roflumilast

INTERVENTIONS:
Drug: metformin
  Other Names: Glucophage tablets
  Arms: metformin
Drug: liraglutide
  Other Names: Victoza injection
  Arms: liraglutide
Drug: roflumilast
  Other Names: Daxas 500 micrograms film-coated tablets
  Arms: roflumilast

SUMMARY:
The purpose of this study was to determine whether monotherapy treatment with phosphodiesterase-4 (PDE-4) inhibitor roflumilast is more effective than treatment with glucagon-like protein 1 (GLP-1) liraglutide or treatment with metformin as monotherapy in the treatment of obese women with polycystic ovary syndrome (PCOS) regarding weight reduction who have not been treated before. The investigators anticipated greater changes in body weight in patients on roflumilast treatment than in liraglutide or metformin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30 kg/m² or higher

Exclusion Criteria:

* depression
* type 1 or type 2 diabetes mellitus
* history of carcinoma
* history of pancreatitis
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* significant cardiovascular, kidney or hepatic disease
* the use of medications other than metformin known or suspected to affect reproductive or metabolic functions
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in body weight. | Patient's body weight was mesured at the base point and every four weeks during 12 weeks of clinical trial.
  The patient's body weight was measured in kilograms.

SECONDARY OUTCOMES:
The secondary outcome was change in body mass index (BMI). | Patient's body weight were measured at the basepoint and every four weeks during the 12 weeks of clinical trial. Patient's height was measured at the basepoint.
  Patient's BMI was defined as the patient's body mass in kilograms divided by the square of their height in meters.
The secondary outcome was change in waist circumference. | Patient's waist circumference was measured at the basepoint and every four weeks during 12 weeks of clinical trial.
  Patient's waist circumference was measured in centimeters.

OTHER OUTCOMES:
The other outcomes was changes in fasting concentrations of glucose. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
Other outcome was change in fasting concentration of insulin. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Fasting concentrations of insulin was measured in mU/L.
Other outcome was change in blood concentrations of LH (luteinizing hormone). | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentration of LH was measured in U/L.
Other outcome was change in blood concentrations of FSH (follicle-stimulating hormone). | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of FSH was measured in U/L.
Other outcome was change in blood concentration of testosterone. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentration was measured in nmol/L.
Other outcome was change in blood concentration in androstenedione. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of androstenedione was measured in nmol/L.
Other outcome was change in blood concentrations of SHBG (sex hormone-binding globulin). | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of SHBG was measured in nmol/L.
Other outcome was change in blood concentration of DHEAS (dehydroepiandrosterone sulfate). | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of DHEAS was measured in micromol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Jensterle M, Salamun V, Kocjan T, Vrtacnik Bokal E, Janez A. Short term monotherapy with GLP-1 receptor agonist liraglutide or PDE 4 inhibitor roflumilast is superior to metformin in weight loss in obese PCOS women: a pilot randomized study. J Ovarian Res. 2015 Jun 2;8:32. doi: 10.1186/s13048-015-0161-3. PMID 26032655